CLINICAL TRIAL: NCT00555425
Title: Buprenorphine Maintenance vs. Detoxification in Prescription Opioid Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0504027597; 1R01DA020576-01A1 (NIH); R01DA020576 (NIH); DPMC (Other: NIDA); NCT00595400 (obsolete NCT alias)
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Opiate Dependence
Keywords: Buprenorphine; Buprenorphine/naloxone; Counseling; Primary care
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Buprenorphine/naloxone maintenance (Mtn) is designed to reflect usual care by primary care physicians and includes weekly drug counseling (DC) and referral to ancillary services.
  Interventions: Behavioral: Behavioral: Buprenorphine/naloxone maintenance (Mtn)
- 2 (Experimental): Buprenorphine/naloxone detoxification (Dtx) is identical to Mtn for the first 4 weeks (stabilization) following randomization. In Mtn, Bup will continue unchanged for the remainder of the study. In Dtx, the dosage of Bup will be tapered to zero over the next 3 weeks, and patients will not receive additional Bup for the remainder of the study. Dtx patients will be offered thrice-weekly DC beginning during the taper and naltrexone will be offered 7 days following the last dose of Buprenorphine/naloxone.
  Interventions: Behavioral: Behavioral: Buprenorphine/naloxone detoxification (Dtx)

INTERVENTIONS:
Behavioral: Behavioral: Buprenorphine/naloxone maintenance (Mtn) — Mtn is designed to reflect usual care by primary care physicians and includes weekly drug counseling (DC) and referral to ancillary services. Dtx and Mtn will be identical for the first 4 weeks (stabilization) following randomization. In Mtn, Bup will continue unchanged for the remainder of the study.
  Arms: 1
Behavioral: Behavioral: Buprenorphine/naloxone detoxification (Dtx) — Dtx and Mtn will be identical for the first 4 weeks (stabilization) following randomization. In Dtx, the dosage of Bup will be tapered to zero over the next 3 weeks, and patients will not receive additional Bup for the remainder of the study. Dtx patients will be offered thrice-weekly DC beginning during the taper and naltrexone will be offered 7 days following the last dose of Bup.
  Arms: 2

SUMMARY:
The aim of the study is to determine whether buprenorphine/naloxone maintenance versus detoxification using buprenorphine/naloxone, in prescription opioid dependent patients receiving primary care management and drug counseling in an office-based setting, leads to decreased illicit opioid use.

DETAILED DESCRIPTION:
Prescription opioid dependence is increasing and creates a significant public health burden, but office-based physicians lack evidence-based guidelines to decide between maintenance or detoxification treatment with buprenorphine/naloxone. The proposed study compares buprenorphine/naloxone maintenance (Mtn) vs. detoxification (Dtx) in a 18-week randomized clinical trail in a heterogeneous population of prescription opioid dependent patients (N=120) in a primary care clinic. Patients are randomized to Mtn or Dtx after a 2-week induction period. Mtn is designed to reflect usual care by primary care physicians and includes weekly drug counseling (DC) and referral to ancillary services. Dtx and Mtn will be identical for the first 4 weeks (stabilization) following randomization. In Mtn, buprenorphine/naloxone will continue unchanged for the remainder of the study. In Dtx, the dosage of buprenorphine/naloxone will be tapered to zero over the next 3 weeks, and patients will not receive additional buprenorphine/naloxone for the remainder of the study. Dtx patients will be offered thrice-weekly DC beginning during the taper and naltrexone will be offered 7 days following the last dose of Bup. The study will test the hypothesis that Mtn will lead to decreased illicit drug use and will demonstrate incremental cost-effectiveness compared to Dtx. Relevance to public health: The results of this study will help define the role of maintenance vs. detoxification with buprenorphine/naloxone in the care of prescription opioid dependent patients in primary care.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence

Exclusion Criteria:

* current dependence on alcohol, cocaine, benzodiazepines or sedatives
* current suicide or homicide risk
* current psychotic disorder or untreated major depression
* inability to read or understand English
* life-threatening or unstable medical problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Fiellin, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - The APT Foundation, Inc. -- Welch Building, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

REFERENCES:
- [Derived] Fiellin DA, Schottenfeld RS, Cutter CJ, Moore BA, Barry DT, O'Connor PG. Primary care-based buprenorphine taper vs maintenance therapy for prescription opioid dependence: a randomized clinical trial. JAMA Intern Med. 2014 Dec;174(12):1947-54. doi: 10.1001/jamainternmed.2014.5302. PMID 25330017

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 289 Patients underwent assessment for eligibility, 29 did not meet inclusion criteria, 132 lost contact or chose other treatment, and 15 did not complete induction
Groups:
- Taper Condition: Buprenorphine/naloxone detoxification (Dtx) is identical to Mtn for the first 4 weeks (stabilization) following randomization. In Mtn, Bup will continue unchanged for the remainder of the study. In Dtx, the dosage of Bup will be tapered to zero over the next 3 weeks, and patients will not receive additional Bup for the remainder of the study. Dtx patients will be offered thrice-weekly DC beginning during the taper and naltrexone will be offered 7 days following the last dose of Buprenorphine/naloxone.
  Behavioral: Buprenorphine/naloxone detoxification (Dtx): Dtx and Mtn will be identical for the first 4 weeks (stabilization) following randomization. In Dtx, the dosage of Bup will be tapered to zero over the next 3 weeks, and patients will not receive additional Bup for the remainder of the study. Dtx patients will be offered thrice-weekly DC beginning during the taper and naltrexone will be offered 7 days following the last dose of Bup.
- Maintenance Condition: Buprenorphine/naloxone maintenance (Mtn) is designed to reflect usual care by primary care physicians and includes weekly drug counseling (DC) and referral to ancillary services.
  Behavioral: Buprenorphine/naloxone maintenance (Mtn): Mtn is designed to reflect usual care by primary care physicians and includes weekly drug counseling (DC) and referral to ancillary services. Dtx and Mtn will be identical for the first 4 weeks (stabilization) following randomization. In Mtn, Bup will continue unchanged for the remainder of the study.
Period: Overall Study
Arm/Group | Taper Condition | Maintenance Condition
Started | 57 | 56
Completed | 6 | 37
Not Completed | 51 | 19
Not completed — Missed Medication > 1 wk | 34 | 15
Not completed — Missed 3 physician management visits | 1 | 0
Not completed — Met criteria for protective transfer | 16 | 3
Not completed — Became pregnant and transferred care | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Taper Condition | Maintenance Condition | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (8.8) | 30.5 (9.8) | 30.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 34 | 31 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 53 | 52 | 105
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 56 | 52 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Illicit Opioid Use
Description: Urinalysis based on scheduled weekly urine screenings during treatment period
Time Frame: 18 weeks
Measure: Mean (95% Confidence Interval); unit: percent of opioid negative urine samples
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 57 | 56
percent of opioid negative urine samples | 35.2 [26.2 to 44.2] | 53.2 [44.3 to 62.0]

2. Secondary Outcome: Proportion of Patients Protectively Transferred
Description: >= 2 consecutive weeks of daily illicit opioid use and opioid positive urine samples after completion of the first 6 weeks of the study
Time Frame: 18 weeks
Measure: Number; unit: participants
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 57 | 56
participants | 16 | 3

3. Secondary Outcome: Retention in Treatment
Description: Mean number of days from randomization to last clinical contact
Time Frame: 18 weeks
Measure: Mean (95% Confidence Interval); unit: number of days
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 57 | 56
number of days | 57.5 [47.0 to 59.9] | 98.7 [88 to 109.4]

4. Secondary Outcome: Reduction in Cocaine Use
Description: As measured by the percent of provided urines positive for cocaine
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: percent of cocaine positive urines
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 57 | 56
percent of cocaine positive urines | 11.5 (25.9) | 11.1 (23.5)

5. Secondary Outcome: Changes in HIV Risk
Description: As measured by the AIDS Risk Inventory. The AIDS Risk Inventory (ARI) is a 166 item structured interview that assesses the number and frequency of drug-related and sexual risk behaviors in the preceding 3 months. Calculation of the ARI total score is based on the frequency of occurrence of a given behavior and on the recency of this behavior, with recency being weighted more than a life-time occurrence of the same behavior. Higher values are associated with greater risk of HIV transmission (worse).
  There are 10 subscales comprised of between 8 and 24 items. Subscales scores are based on the sum of the individual items and the overall ARI total score is the sum of the subscales.
  Scores can range from 0 to 350, although among opioid dependent patients most values are below 100 with means between 50 and 60 depending on characteristics of the patients and treatment status.
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 57 | 56
units on a scale
  Baseline | 66.7 (25.6) | 67.6 (25.7)
  18 weeks | 74.5 (19.4) | 74.4 (18)

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction as measured by survey. Primary Care Buprenorphine Satisfaction Scale (PCBSS). Comprises of 19 items evaluating satisfaction with staff expertise, concern, and responsiveness. Range of scores from 15-95. I higher score indicates greater satisfaction.
Time Frame: 18 weeks
Population: Results are provided on those individuals who completed this assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 37 | 45
units on a scale | 78.7 [73.9 to 83.4] | 79.9 [75.2 to 84.7]

7. Secondary Outcome: Health Status
Description: Measured by the SF-36 overall transformed measure. In the SF-36 all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: 18 weeks
Population: Results are provided on those individuals who completed this assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taper Condition | Maintenance Condition
Number analyzed (Participants) | 47 | 54
units on a scale
  Baseline | 67.2 (20.4) | 67.6 (18.6)
  In-Treatment | 68.7 (30.5) | 66.6 (21.9)

ADVERSE EVENTS:
Arm/Group | Taper Condition | Maintenance Condition
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No